#### **LEGAL GUARDIAN CONSENT FORM**

## **LEGAL GUARDIAN CONSENT FORM FOR SCREENING AND ENROLMENT**

**Study Title:** A Demonstration Open Label Study to Assess the Acceptability and Use of Truvada Pre-exposure Prophylaxis in Healthy, HIV-Uninfected Adolescents, 15-19 Years of Age.

**Study Number: DAIDS ES ID 11931** 

**Study Sponsor: Desmond Tutu HIV Foundation** 

Principal Investigator Prof Linda-Gail Bekker

Site Address Desmond Tutu HIV Foundation

**Guinea Fowl Road** 

Masiphumelele

Site Telephone Number 021 785 5454

To the potential participant: This consent form may contain words that you do not understand. To help you understand these words we have included simpler words in brackets after complex ones. Please ask the study doctor or the study staff to explain any words or information that you do not clearly understand. You may take home an unsigned copy of this consent form to think about or discuss with family or friends before making your decision.

## **INTRODUCTION**

The Desmond Tutu HIV Foundation is doing a study of young people and a medication called Truvada, and you and your child are being invited to take part.

Before agreeing to be screened for enrolment into the study, it is important that you read and understand the following explanation of the purpose (reason for) of the study, the study procedures (what will happen during the study), benefits, risks, and you and your child's right to withdraw from the study at any time.

This form has information to help you decide if you want your child to participate. If you decide for your child to take part you will sign this form because your child is younger than 18 years. Your child will also need to sign a form. If your child turns 18 while she/he is participating in the study she/he will sign another form because she/he will be able to consent without your permission.

## **ABOUT THE STUDY**

South African adolescents are at risk for HIV infection. Rates of HIV infection, mostly through sexual transmission, among adolescents are increasing rapidly. Therefore, prevention methods to lower HIV risk among adolescents are urgently needed.

This is part of a bigger project called The CHAMPS (Choices for HIV Adolescent Methods of Prevention in South Africa) project. In this project we are assessing whether an HIV prevention "menu" can be developed for adolescents in South Africa. What we mean by this is that it may mean that people can apply different prevention tools to their lives, e.g. Condoms as well as PrEP. The CHAMPS project is comprised of three pilot studies rolled out as a series of small, focused, interrelated protocols and will help us understand how your child may choose to use various prevention tools when they know what tools are on offer.

The purpose of this research study is to find out whether adolescents will use the medication called Truvada as an HIV prevention tool. Truvada is a type of antiretroviral (ARV) medication that is commonly used to treat HIV when used in combination with another drug. Truvada is not effective when used alone in the treatment of HIV infection in HIV positive individuals. Truvada is now also being tested as a pre-exposure prophylaxis or PrEP. PrEP is an experimental approach

Protocol CHAMPS PlusPills Version 1.0 dated June 2014 Approved by University of Cape Town Human Research Ethics Committee on 11/Aug/2014

English Legal Guardian Consent Form for Screening and Enrolment Version 3.0 dated 24 July 2015

that uses ARVs to prevent HIV infection in HIV-negative people—it is used by HIV negative persons to protect them against possible infection with HIV.

We do not know the effects of PrEP in adolescents between the ages of 15 and 19 years, and we do not know if it protects adolescents from getting HIV. Because of this, the South African Medicines Control Council (MCC) has not yet approved Truvada for preventing HIV infection in adolescents. The MCC however, has given permission for a study to be conducted to establish how safe it is for adolescents to use Truvada and whether they would find it acceptable to use the medication as instructed.

A number of studies have been conducted to show that Truvada is safe in HIV uninfected men and women over 18 years of age. Four studies, whose results were announced in 2010, 2011 and 2013, showed that HIV infection among adult men and women can be prevented by taking Truvada daily. These adult studies involved adult males and females, men who have sex with men (in South Africa) and sero-discordant couples (where one partner is HIV positive and the other is HIV negative) as well as people who inject drugs. Adult studies have shown that even though the risk of HIV was reduced, HIV infections still occurred. We do not know whether it is safe yet nor can we say whether it can stop some HIV infections in adolescents between the ages of 15 and 19 years.

We will enroll 75 adolescents aged 15 to 19 years at the Masiphumelele Clinic in Cape Town and 75 adolescents at the Perinatal HIV Research Unit (PHRU) site which is based in Kliptown, located near Soweto, close to Johannesburg. We want to answer several questions during the study:

- Will adolescents use the study medication (Truvada) in the way in which they have been told to take it?
- What helps young people adhere to, or keep taking, the study medication?
- How do young people's relationships, attitudes, and sexual behaviour change over time, while taking this medication?

• Is the study medication (Truvada) safe for young people 15-19 years old?

To see if your child can join this study, there are a number of screening procedures we need to do. These include:

- Interview questions
- Urine tests
- Blood tests
- Physical examination

Your child can **not** participate in this study if they are:

- HIV positive
- Hepatitis B positive
- Currently taking part in another HIV prevention study that involves medication
- (For females) Pregnant or planning on becoming pregnant or breastfeeding
- Has a job or other obligations that would require long absences from the area (> 4 weeks at a time)

### **SCREENING PROCEDURES**

In order to find out if your child is eligible to participate in the study, you and your child will be asked to consent to some screening tests, once they are fully explained to both of you. These tests may take more than one visit and may take 1-2 hours to complete. All screening tests must be done within 40 days. If all tests are not done within 40 days, and you and your child still want to find out if your child is eligible for the study, you will both have to be re-consented and your child must begin the screening tests again.

The following procedures will occur at the screening visit:

• An identification number will be assigned to your child.

- Your child will be counseled about HIV before having an HIV test. We will
  take some blood from your child's finger (about a drop) for the HIV test.
  Your child will be told their result as soon as it is available at this visit.
  Your child will talk with the study staff about the meaning of their result
  and how they feel about it.
- If the test shows that your child has HIV, they cannot continue with the screening nor take part in the study. Your child will receive counseling and referral for HIV care and treatment. Your child will be encouraged to share their results with an adult whom they trust. If their test results show that your child does not have HIV, they may continue with the screening.
- A trained medical staff member will conduct a full physical examination of your child.
- Your child will also need to answer questions about themself, which will
  include where they live, their health and medical history, and personal
  questions about their relationships and sexual behaviour. Your child
  cannot take part in this study if they are not sexually active. You will
  therefore be aware that your child is sexually active if they do take part.
- If your child is female, the study doctor and/or study nurse will ask your child to give some urine for a pregnancy test. Your daughter will be required to take a low dose hormonal birth control (the pill or injection) during the study, which we will provide. She can receive information about contraception and access to contraceptives without your consent, and we will counsel her to practice safer sex. If she is pregnant, she cannot take part in the study. We will not tell you but will encourage her to tell an adult she can trust. We will counsel her about her options in relation to her pregnancy.

- We will take one tube, about 5 mls (about 1 teaspoon) of blood with a
  needle from your child's arm to check how well their kidneys and liver
  are working as well as checking their general health.
- We will take two tubes, about 10 mls (about 2 teaspoons) of blood to check for Hepatitis B infection. Hepatitis B is a virus that causes inflammation of the liver. This infection is spread in a similar way as the HIV virus, that is, from mother to child, through contaminated blood, and in some cases through sexual transmission. Tenofovir, one of the active ingredients in the study medication, can be used to treat both Hepatitis B and HIV. The blood will be sent to a laboratory for testing and your child will be provided with their test results. If we find that your child has Hepatitis B infection, they may not participate in the study. Your child will receive appropriate counselling and referrals. If we find that your child does not have Hepatitis B infection, the study staff will vaccinate your child (give your child three separate injections) that will prevent this disease in the future.
- Your child will be tested for, and counseled about, other infections that
  may be passed on to them during sex, including herpes (HSV-2),
  chlamydia, and gonorrhea, which are sexually transmitted infections
  (STIs). If your child is having health problems that may be due to these
  infections, we will help them get the appropriate medical care.
  - Chlamydia, and gonorrhea are bacterial infections. If a person takes medicines, they will go away completely. We will test your child for chlamydia and gonorrhea at screening, at Month 3, and at their final study visit.
  - Herpes is a virus which may cause painful sores in the genital area.
     However, herpes may cause no symptoms at all. If painful sores
     from herpes arise, they can be treated with medicine. The herpes

virus always stays with a person and may be spread to their sexual partners. We will test your child for herpes at screening, month 3 and at their final study visit. If you child has sores, we will help them get medicine to help the sores go away.

- Your child will be asked about medications they are currently taking, previous medical problems they may have had, and will have a physical examination. Your child should be open with their study doctor or study nurse regarding their health history, since by not disclosing all the information about their health, they may put themselves at risk by participating in this study. They will be given appropriate feedback and access to care, should these procedures reveal important information about their health.
- If all the tests show that your child is eligible to participate in the study, we will explain the study to you and your child again and check that you both are still willing for your child to continue in the study and answer any questions you have.
- Your child may be given a vaccine injection to protect against Hepatitis B, if they have not been previously vaccinated.
- If you and your child are in agreement and decide for your child to be enrolled in the study, you will be asked to sign this document to confirm your understanding of and participation in the study. You will be given a copy of this Guardian Consent Form for Screening and Enrolment Version 3.0 dated 24 July 2015 to keep.
- After reading this document, the study doctor and/or study nurse will ask your child to complete a short quiz in order to make sure that you understand what you have consented to for enrolment. If your child gets enough of the answers right, your child will be able to continue with enrolment. Your child has three chances for this. If after three chances your child has still not got enough answers right, your child will not be

- able to continue in the study. This is to make sure that you are making an informed decision about taking part.
- Both you and your child need to be in agreement in order for your child to
  be enrolled. Your child will also be asked to read or will have an
  information form read to them. If they agree, they will be asked to sign a
  copy and will be given a copy to take home. You will also need to
  complete the test to ensure that you understand what you are consenting
  to when your child takes part in the study.
- Even though you must give consent for your child to be enrolled in the study, your child will be giving their own assent to take part and will consent independently for tests that we will perform and treatment that she/he may receive during the study. We will tell you more about these tests in the next sections.
- Your child's decision to continue in the study or to withdraw will not
  affect your child's regular care or harm your child's relationship with the
  study doctor and/or study nurse.

## **ENROLMENT VISIT**

This visit may take about 3 hours to complete. In addition to the above procedures, the following will happen:

- Study staff will provide your child with any test results received since the screening visit(s).
- Study staff will ask your child to provide information on their health history and any medical events that have taken place since the screening visit.
- Study staff will take some blood from your child's finger (about a drop)
  for the HIV test. Your child will be told their result as soon as it is
  available at this visit. Your child will receive pre- and post-test counseling,
  which will include risk reduction counseling.

- Female participants will be asked to give some urine at each visit for a
  pregnancy test. Study staff will talk with your child about her choices and
  will ask about her use of contraception at each study visit.
- Your child will also need to answer personal questions about their relationships, attitudes, and sexual behaviour.
- Study staff will ask your child to update the information on where you live and on how they can keep in contact with you and your child.
- We will provide your child with enough condoms until the next study visit and discuss how to use them and how your child can protect himself/herself from becoming infected with HIV.
- Your child may be given a vaccine injection to protect against Hepatitis B, if they have not been previously vaccinated.
- Your child will be asked to take the study medication "Truvada" one pill every day of the week for the next month. They will be given enough pills for 30 days.
- Your child will be counseled about the need for adherence. Throughout the study your child will also have blood taken to test how much Truvada there actually is in your child's blood. This result will be available at the next study visit. Your child will be asked whether he/she wishes to receive this result or whether they prefer to be counseled without this result. Research staff will give the results and counsel your child accordingly. Those who choose not to get these results will still receive standard counseling on how and why they should take the pills.

#### **FOLLOW-UP VISITS**

Your child will complete monthly follow-up visits (approximately every 30 days) during the first three months of the study, after he/she enrols. These follow-up visits will take about 60 to 90 minutes and the following will occur:

- Study staff will take some blood from your child's finger (about a drop)
  for the HIV test. Your child will be told their result as soon as it is
  available at this visit. Your child will talk with the study staff about the
  meaning of their result and how they feel about it. Your child will receive
  pre- and post-test counseling, which will include risk reduction
  counseling.
- Female participants will be asked to give some urine at each visit for a
  pregnancy test. If your daughter becomes pregnant, it is necessary that
  she stops using the medication. Study staff will talk with your child about
  her choices and will ask about her use of contraception at each study visit.
- Your child will also need to answer personal questions about their relationships, attitudes, and sexual behaviour.
- Study staff will ask your child to update the information on where they live and on how staff can keep in contact with both of you.
- We will provide your child with enough condoms until the next study visit and discuss how to use them and how they can protect themselves from becoming infected with HIV.
- Should your child have any symptoms that cause concern, they will be asked to have a physical examination. Every 3 months, your child will receive a full physical examination.
- Your child will be given study medication (Truvada) and asked to take a pill a day every day until the next scheduled visit. They will be re-issued with medication at every scheduled visit for 3 months.
- Study staff will ask your child about how well they have taken the medication and any side effects or difficulties that may have occurred.
- Study staff will also collect some blood, approximately 5 mls (1 teaspoon)
  from your child to check their general health and to determine the
  amount of study medication in their blood. Results from some of these

blood tests will be given to participants who wish to hear these results, in order for the research team to understand if that affects their usage of the study medication.

## **FOLLOW-UP VISITS (MONTHS 4-12)**

At the 3-month visit, your child will be offered study medication, but will be allowed to choose whether they prefer to continue with it or stop it. It is your child's choice whether or not to take this medication. Your child may decide that they do not want to take study medication, or your child may choose to take the study medication at a later time. Your child will be asked about their choice every 3 months by the study staff.

If your child chooses not to take the study medication at any time, your child can still remain in the study and will be asked to attend all visits.

At the end of month 3, your child will begin 3 monthly visits, approximately every 90 days for the remaining 9 months.

Participants will receive blood tests throughout the study that measure the amount of study medication in their blood. These tests are called Dried Blood Spots and involve pricking your child's vein, taking a small amount of their blood, and drying a blood spot on a special piece of paper. These tests will occur at all study visits, and at the next visit, your child will be shown the result of the test if they wish to receive this – it is their choice. Either way, they will be counseled about the use of the Truvada pills.

For study participants who agree to take the study medication, the following procedures will also be conducted during follow up visits during Month 4-12:

Study staff will take some blood from your child's finger (about a drop)
for the HIV test. Your child will be told their result as soon as it is
available at this visit. Your child will talk with the study staff about the
meaning of their result and how they feel about it. Your child will receive
pre- and post-test counseling, which will include risk reduction
counseling.

- Your child will have urine testing
- Female participants will be asked to give some urine at each visit for a
  pregnancy test. If your child becomes pregnant, it is necessary that she
  stops using the medication. Study staff will talk with her about her
  choices and will ask about her use of contraception at each study visit.
- Your child will also need to answer personal questions about their relationships, attitudes, and sexual behaviour.
- Study staff will ask your child to update the information on where they live and on how they can keep in contact with your child.
- Your child will be given enough study medication until the next study visit and instructed about how to take it.
- We will remind your child to use their study medication daily by SMS (if they choose to receive it) and ask your child if they are experiencing any problems using the medication.
- Your child must bring back all unused study medication to the study staff.
- We will provide your child with enough condoms until the next study visit and discuss how to use them and how your child can protect themselves from becoming infected with HIV.
- Should your child have any symptoms that cause concern, they will be
  asked to have a physical examination. For the rest of the study, your child
  will receive a full physical examination every 3 months.
- Study staff will also collect some blood, approximately 5 mls (1 teaspoon) to check your child's general health and to determine the amount of study medication in their blood. Results from some of these blood tests will be given to those who wish, in order for the research team to understand if that affects their usage of the study medication.

- Every three months, your child will be asked by a study staff member again about whether or not h/she wishes to take the study medication.
   Your child can either stop or start the study medication at these visits.
- At each adherence counseling session your child will be asked whether
  they wish to receive blood drug level results. This is voluntary. We will
  ask your child why he/she has made the choice they do.
- Your child will be asked about any social harms or benefits they have experienced as a result of participating in the study.

## **SECOND FINAL STUDY VISIT**

## These procedures will also be done at an early discontinuation visit

- Your child's second final study visit will be at Month 12 (Week 48).
- Study staff will take some blood from your child's finger (about a drop)
   for the HIV test. You child will be told their result as soon as it is available at this visit.
- Urine testing in your child will be performed.
- Female participants will be asked to give some urine at each visit for a pregnancy test.
- Study staff will test your child for herpes (HSV-2), chlamydia, and gonorrhea.
- Study staff will ask your child personal questions about their relationships, attitudes, sexual behavior, and opinions about the study medication.
- Study staff will also collect some blood, approximately 5 mls (1 teaspoon)
  to check your child's general health and to determine the amount of study
  medication in their blood.

## **FINAL STUDY VISIT (week 52)**

- Study staff will ask your child some personal questions about your child's relationships, attitudes, sexual behavior and opinions about the study medication.
- All final and outstanding blood results will be returned.

### **FOCUS GROUPS**

 Between Month 11 and 12, some participants will be randomly selected to attend a focus discussion group about their experiences with taking the medication, their likes, dislikes, where they would like to access it if it is licensed and how they think they would use it. Your child may be asked to participate. This is voluntary – your child may decline.

## **LEAVING THE STUDY**

Tell us if you or your child decides to leave the study or if your child stops taking the medication.

You and/or your child are free to leave/withdraw consent from the study at any time and for any reason. Your child's care at this clinic and their legal rights will not be affected, but it is important for you to let us know.

We will ask your child to come back to the clinic one last time. We may ask to take some blood and urine samples. We will also ask about any personal problems or benefits your child has experienced from being in the study and ask them to complete a questionnaire about why they want to leave the study.

## IF YOUR CHILD BECOMES INFECTED WITH HIV DURING THIS STUDY

It is important to identify people with HIV early so that they can get the services that they need.

If the HIV test result is positive, your child will receive counseling from study staff. They will be encouraged to share their test results with an adult they trust. This does not have to be their parent/legal guardian. Your child will also be referred for appropriate care and support services in the community. Your child may be asked to join other studies that may be going on at this study clinic.

Following another pretest information session, a blood sample for CD4 count will be obtained. These tests will provide the doctor with more information about their health, immunity, and the nature of the disease. When your child returns to the clinic for the next interim visit, results of the CD4 count will be discussed and a referral letter to a Primary Health Care facility will be prepared. Your child will be followed up for one year beyond sero-conversion and will have a CD4 at 3 monthly intervals to ensure that initial care is well-managed.

If your child becomes infected with HIV during this study, and this has been confirmed with the procedures described above, your child will be told to stop using the study medication because we are not sure about the effects of the study medication in HIV infected people. Your child will be invited to continue with the remainder of the study visits, and will be supported with disclosure to a trusted adult. A genotype test will be performed on the HIV Virus from your child's blood to help with management.

#### **AT ANY TIME DURING THE STUDY**

Your child will be asked to tell the study staff about medical problems your child may have during the study. You or your child can also contact the study staff between regular visits to report these problems. The study staff will examine your child as needed and will either provide or refer your child for medical care that they may need.

If your child is having health problems that may be caused by infections passed during sex, they will be given a physical examination. Your child will get treatment for curable infections passed on to them during sex if they need it. If your child has any infections that their partner may also have, they can bring him or her to the trial site for treatment that may be needed. This will be at no cost to them or their partner.

Your child can have extra counseling and testing for HIV if needed between regular visits. If they wish, their partner can have HIV counseling and testing with them.

Your child or the study staff may request an interim study visit at any time.

During this study your child may also be asked to participate in other sub-studies (studies related to this one). Your child does not have to participate in any substudies if they do not want to. You and your child will be given as parate consent to sign for each sub-study that they wish to participate in.

While your child is in this study, we ask that they please:

- Do not share their study medication with anyone else or use study medication that doesn't belong to them.
- Do not participate in any other study involving other HIV prevention medication - this is important for their own safety:
  - If your child uses other study medication from different studies at the same time and then has a problem that requires medical attention, we will not know which medication has caused the problem.
  - If your child is using study medication from different studies at the same time, we cannot assess which study medication is working.
- Remember that the medication that we are testing has not been proven
  for safety in adolescents and we do not know if it can prevent HIV
  infection, so it is important that your child continues to use male and
  female condoms, and engages in other safer sex behaviours.

#### **CONTACT**

Once you and your child join the study, it is very important for us to stay in touch with you and find out how you and your child are doing. We will ask for your name, address, phone number, and other contact information at your child's first study visit. We also will ask for the names and contact information of people whom we may contact if we cannot reach you.

We will ask your child to update this information at each study visit. We will use your contact information to remind your child of scheduled study visits. If your

child misses a visit, we may call you with your permission or send letters or visit your home to find you and your child. We will also try to reach you through the contact people that you list for us. If we talk to these people, we will not tell them why we are trying to reach your child.

### RISKS AND/OR DISCOMFORTS OF STUDY PARTICIPATION

#### Risks of blood draws:

In this study, we will take some blood samples. Blood draws can cause bruising, pain, fainting, soreness, redness, swelling, itching, and (rarely) infection where the needle was put in.

## Personal problems/discrimination:

Some participants report personal problems or discrimination because of being in a study. This could happen to your child. Family or friends may worry, get upset or angry, or assume that your child is infected with HIV and treat them badly as a result. If you or your child has bad things happen because of the study, please tell us. We will try to help.

## **Embarrassment/anxiety:**

Your child may feel embarrassed when we ask personal questions about relationships, attitudes, and sex. Your child may feel nervous or scared waiting for their study test results. Your child could feel worried if their test results show that they are infected with HIV, herpes, chlamydia or gonorrhoea. If they are feeling this way, we will try to help her / him feel better.

## Risks of someone finding out your personal information:

We will protect you and your child's personal information. The risk of someone seeing your child's personal information, when they should not have done so, is very low. However, if that happened, you both could feel upset and embarrassed. Someone could use the information to treat you and your child badly. We can tell you more about how we will protect your personal information if you would like it.

## Side effects from the study medication:

Your child may have side effects from taking the study medication. The most common risks and side effects from the study drug include dizziness, fatigue, difficulty sleeping, depression, strange dreams, diarrhea, nausea (upset

stomach), vomiting, headache, rash and gas. Skin discoloration (small spots or freckles) may also occur.

Less common but more serious risks may include:

- Liver problems
- Kidney problems
- Inflammation of the pancreas
- Anemia (low red blood cells)
- Lactic acidosis (a buildup of a chemical called lactate in the body that can cause symptoms of unexplained weight loss, stomach discomfort, nausea, vomiting, fatigue, cramps, muscle pain, weakness and shortness of breath)
- Lipodystrophy (changes in fat distribution in your body such as an increase in fat around the waist, back of the neck and breast areas, and thinning of the face, legs and arms)
- Metabolic disorders (changes to lipid and sugar levels in your blood)
- Changes in bone mineral density (thinning bones). This may be made
  worse if your child is also using injectable hormonal methods of family
  planning, e.g. nur isterate IMI.
- Allergic reactions (symptoms may include fever, rash, upset stomach, vomiting, loose or watery stools, abdominal pain, achiness, shortness of breath, a general feeling of illness or a potentially serious swelling of the face, lips, and/or tongue;
- If your child is infected with hepatitis B virus, flare-ups of this infection
  may occur. We will minimise this risk by screening your child for
  Hepatitis B and vaccinating them if they are not yet vaccinated or
  infected.

- Resistance: if your child becomes infected with HIV and is taking Truvada,
  there is a risk that the HIV virus in your child's blood may change its make
  up and become resistant to this antiretroviral medication. This means
  your child would not be able to use this medication for treatment of their
  HIV. We will try to minimise this risk by making sure your child is not HIV
  infected when s/he starts the treatment and also by testing her / him for
  HIV frequently.
- The study medication is investigational (experimental) and there may be other risks or side effects which are unforeseen or unknown. You or your child should immediately contact the study doctor or study nurse if any side effects occur throughout their participation in this study.

We will try to minimize any side effects and/or risks to your child's safety and well-being. Tests will be done to carefully monitor your child's physical and mental health, including their kidney and liver functioning. The study doctor or study nurse will ask your child about any side effects they have experienced at every visit and a full physical exam will be conducted as needed or every 3 months. Your child will be provided with information about how to prevent HIV and will have access to counseling, support, and other social and health-related services as needed.

## EARLY TERMINATION/DISCONTINUATION

There are some situations where we would need to stop your child from taking Truvada. These are as follows:

- Toxicity related to Truvada
- Your child needs to take medication that cannot be taken while they are taking Truvada
- Your child becomes HIV infected
- Your child is pregnant/breastfeeding
- Your child has completed the study

- Your child has requested to stop taking Truvada
- Any conditions or clinical reasons that will threaten your child's safety and well-being

There are certain situations where we may discontinue your child's participation in the study. These are as follows:

- We are unable to contact your child after a number of attempts
- Your child is repeatedly not taking Truvada as prescribed
- Your child is pregnant/breastfeeding
- Your child requests to be withdrawn from the study
- You no longer thinks the study is in your child's best interests
- Your child is judged by the Site Investigator to be at significant risk of failing to comply with the provisions of the protocol as to cause harm to him/herself or seriously interfere with the validity of study results
- At the discretion of the Independent Ethics Committee, Medicines Control Council, Site Investigator, or pharmaceutical supporter.
- DAIDS, NIAID, the Office of Human Research Protection (OHRP), and the FDA as regulatory entities may also discontinue the study at their discretion.

## **BENEFITS OF STUDY PARTICIPATION**

- We will give your child condoms and show them how to use them, and
  counsel them on how to prevent HIV, and provide them with referrals for
  male circumcision, Post Exposure Prophylaxis or PEP (a medication that
  someone can take after they might have been exposed to HIV), and
  reminders that STI treatment may assist in the prevention of HIV.
- Your child will have physical examinations and some lab tests over the course of the study. This may help them to identify health problems that they did not know about. If we find medical problems during these

- procedures, we will provide your child with treatment if it is provided at this clinic or we will refer your child to another clinic or services.
- Your child will get counseling and testing for HIV and if they are infected with HIV, they will be referred for medical care, counseling, and other services available to them.
- Your child will receive treatment if they show any symptoms of STIs.
- You and your child's participation in this study will contribute to medical knowledge that may help prevent other adolescents from developing HIV.

## PREGNANCY AND CONTRACEPTION (For female participants only)

The risks of the study medication to an unborn baby are not known. Adolescent girls who are pregnant or breastfeeding may not participate in this study. Adolescent girls who become pregnant during the study will remain in the study but will be instructed to stop using the study medication while they are pregnant. Your child must confirm that they are not pregnant now, and that they do not intend to become pregnant during the study. If your child suspects that they have become pregnant during this research study they must notify the study doctor or study nurse immediately.

#### **ALTERNATIVE TREATMENT/METHODS FOR HIV PREVENTION**

There are no medications proven to prevent HIV infection in adolescents although medical male circumcision has been shown to reduce infection in young men as young as 15 years. The only known way to prevent HIV infection during sex is to use a condom every time you have sex. Treating STI's may also help. It may also help to give someone post-exposure prophylaxis after they might have been exposed to HIV. That is, if there is a chance that they might have been infected with HIV e.g. during rape, they can be treated afterwards with medication. In order for PEP to work, it needs to be taken within 72 hours of becoming exposed.

There may also be other research studies that are testing ways to prevent HIV infection in this area that your child may be eligible for. However, if your child

agrees to participate in an alternative study on HIV prevention that involves an experimental study medication, your child will not be eligible for participation in this study.

### **RIGHTS AS A PARTICIPANT IN THIS STUDY**

Your child's participation in this study is entirely voluntary and your child can refuse to participate, or stop at any time, without stating any reason. Your child's withdrawal will not affect their access to other medical care. If you or your child chooses to withdraw from this study, your child does not waive any of their legal rights as a patient or a research participant at this site. You and your child will be informed of any trial related new information in case it may impact your willingness for your child to participate.

## **COSTS AND REIMBURSEMENT FOR STUDY PARTICIPATION**

You and your child will not be paid for taking part in this study. However the study specific visits, study medication and laboratory tests related to this study will be at no extra cost to you or your child. Your child will however be reimbursed to cover the costs of transport to and from the clinic and to compensate them for time spent at the clinic. This will be R50 per visit. We will not be able to reimburse your child for visits that are not part of the regular visit schedule.

#### **INSURANCE**

The sponsor has taken out insurance from SHA in the event of a trial-related injury, i.e. harm suffered as a result of participation in the trial. The sponsor agrees to pay all reasonable medical expenses in accordance with the Association of the British Pharmaceutical Guidelines (ABPI) in the event of an injury or side-effect resulting directly from your child's participation in the trial. The ABPI guidelines recommend that the sponsor of the study should pay, without you having to prove that the sponsor is at fault, for any injury resulting from your child getting the study medication or from other procedures carried out in accordance with the protocol for this study. The sponsor will not be liable for any

loss, injuries and/or harm that your child may sustain where the loss is caused by the use of unauthorized medicine or substances during the study; any injury that results from your child not following the protocol requirements or the instructions that the study doctor may give your child; any injury that arises from any action or lack of action to deal adequately with a side effect or reaction to the study medication; an injury that results from negligence on your child's part. By agreeing to participate in this study, you do not give up your right to claim compensation for injury where you can prove negligence. In particular, your right to pursue such a claim in a South African court in terms of South African law must be ensured.

You must notify the study doctor or nurse immediately of any complications, side effects and/or injuries during the study and the nature of the expenses to be covered. Contact information is provided below.

The insurance does not cover and the study will not pay for:

- Medical treatment of other injuries or illnesses.
- Injury caused by not following the research protocol
- Per DAIDS policy DWD-POL-CL-02.00, the US NIH does not have a mechanism to provide direct compensation for research-related injury.

## **CONFIDENTIALITY**

We will do our best to protect your child's private information. Your child's study records will be kept secure. We use a code number in place of your child's name on most records. We will not share your child's name unless someone working on or reviewing the study needs to know it. This may include the research staff, ethics committee members, members of the MCC, FDA, study sponsor (NIAID), and other related agencies.

We will keep the information listed below, private and will not share this information with you:

- Your child's attitudes towards sexual behaviour and reasons for staying in the study.
- Your child's answers to questions about sexual behaviour and whether they are having sex.
- Any birth control information we talk about and your child's access to contraceptives if they choose.
- The results of tests (including pregnancy and STIs) and treatment that your child has consented to without the help of an adult.

To protect your child from harm, we will encourage them to tell a trusted adult (not necessarily their parents/legal guardian) about certain situations. We will help and support them when they tell others about these difficult situations:

- If they become pregnant or have a termination of pregnancy.
- If they have a positive HIV test result.

Also, the law requires us to tell authorities if your child is being sexually or physically abused. The law also requires us to report sexual offenses like rape to the authorities. We will tell your child if we are going to inform the authorities.

Furthermore, if your child is in a relationship with someone who is very much older than s/he and who seems to be using your child in an unfair way, the study staff will give your child support and help. They will encourage your child to talk to a trusted adult, so that they might help your child deal with this situation.

## **WHO HAS REVIEWED THE STUDY**

These screening and enrolment procedures are part of an overall study. We sent the protocol for the whole study to the University of Cape Town Human Research Ethics Committee. This is an independent committee established to help protect the rights of research participants at the Desmond Tutu HIV Foundation research sites.

We also sent it to the South African Medicines Control Council. Both these institutes have given their approval for us to run the study.

We are following ethical guidelines when we run this study. These are the South

African Department of Health Clinical Trial Guidelines 2006, and DOH (2004)

and ICH/GCP Guidelines and the Declaration of Helsinki (last updated October

2013). These guidelines recommend ways to protect the welfare of research

participants. Please ask us for a copy of these guidelines if you would like to see

them.

The study doctor does not have any financial or personal interests with this

organisation that may bias his/her actions.

If you want any information regarding your or your child's **rights as a research** 

participant, or complaints regarding this research study, you may contact

Professor Marc Blockman at the University of Cape Town Human Research

Ethics Committee, which is an independent Committee established to help

protect the rights of research participants on telephone number 021 406 6338.

After you have consulted with the study doctor and/or Ethics Committee and if

they have not provided you with answers to your satisfaction, you should write

to the South African Medicines Control Council (MCC) at:

The Registrar

South African Medicines Control Council

Department of Health

Private Bag X828

**PRETORIA** 

0001

Fax: 012 395 9201

Email: gouwsj@health.gov.za and mogobm@health.gov.za

**EMERGENCY CONTACT** 

If your child requires emergency care, or if hospitalisation is required at any time

during the study or up to 30 days after taking the last dose of study medication,

Protocol CHAMPS PlusPills Version 1.0 dated June 2014 Approved by University of Cape Town Human Research Ethics Committee on 11/Aug/2014

English Legal Guardian Consent Form for Screening and Enrolment Version 3.0 dated 24 July 2015

Page **26** of **30** 

please tell the treating doctor that your child is/was enrolled in this research study and that your child's study doctor and/or study nurse must be informed.

If you or your child has questions or problems at any time during your participation in this study, use the following important contacts.

If you have questions about this study or want to leave this study, contact Cleopatra Jaars 021 785 5454.

If your child has any symptoms that you think may be related to this study, contact Katherine Gill 021 785 3121.

If you have questions about your rights as a research participant, or problems or concerns about how you are being treated in this study, contact Linda-Gail Bekker at  $021\ 650\ 6959$ .

# **INFORMED CONSENT/SIGNATURES**

You will be given a signed copy of this Guardian Consent Form for Screening and Enrolment Version 3.0 dated 24 July 2015 to keep.

 I confirm that I have received and read or have had read to me and understood this Guardian Consent Form for Screening and Enrolment Version 3.0 dated 24 July 2015 for this research study and have had the opportunity to discuss the study and ask questions. My questions have been answered to my satisfaction and I have had time to decide whether I wish my child to take part.

 I understand that sections of any of my child's medical notes may be looked at by responsible individuals associated with the study, study monitors, or from Regulatory Authorities where it is relevant to my child taking part in this research study. I give permission for these individuals to have access to my child's records.

- I understand that my child's participation is voluntary and that s/he is free to withdraw at any time without giving any reason, without her / his medical care or legal rights being affected.
- I agree to my data and the results of the study being published and submitted to Desmond Tutu HIV Foundation's offices, the US National Institutes of Health/Division of AIDS, and the South African Medicines Control Council
- I give permission for my child's personal doctor about my child's participation in the study, if applicable
- I authorise the collection, transfer and processing of my child's study data.

## \* FOR ANY IMPARTIAL WITNESS

I have received and read this Guardian Consent Form for Screening and Enrolment Version 3.0 24 July 2015 and any other written information provided to the participant.

I have attended all verbal discussions between the investigator/study coordinator or designee and participant about the study.

By signing, I attest that the information provided was accurately explained to and apparently understood by the participant and that informed consent was freely given.

#### Printed Name of Guardian

English Legal Guardian Consent Form for Screening and Enrolment Version 3.0 dated 24 July 2015

| Guardian Signature | Date and time |
|----------------------------------------|---------------|
| <u>OR</u> | |
| Participant thumbprint | |
| * Printed Name of Witness | |
| * Signature of Witness | Date and time |
| * Printed Name of Person Conducting Co | nsent |
| (If other than Investigator) | |
| Signature of Person Conducting Consent | Date and time |
| (If other than Investigator) | |
| Printed Name of Investigator | |
| Signature of Investigator | Date and time |

I hereby verify that consent was obtained from the above mentioned person. The participant's guardian has been informed about the risks and the benefits of this study, understands the risks and benefits and gave consent for their child to participate without coercion, undue influence or inappropriate incentives.